CLINICAL TRIAL: NCT05517707
Title: Gravitas Feeding Tube System Placement in Neonates
Status: Completed | Type: Observational
Sponsor: Gravitas Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD-04-1493
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Nasogastric Tube
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Nasogastric tube group: Neonates age 0-18 weeks post-partum at enrollment with gestational age > 28 weeks will have the Gravitas Feeding Tube placed using standard technique. Tube placement will be verified by the institution standard of care. Study tubes are to remain in place up to 30 days.
  Interventions: Device: Nasogastric Tube

INTERVENTIONS:
Device: Nasogastric Tube — Temperature and impedance data will be collected from sensors embedded within the feeding tube wall.

SUMMARY:
The purpose of this study is to optimize the Gravitas Feeding Tube System Placement Algorithm for NICU patients and to evaluate the safety and effectiveness of the Gravitas Feeding Tube in the neonate population for the administration of nutrition, fluids and medications.

ELIGIBILITY:
Infants in the Newborn Intensive Care Unit requiring a 5Fr NG tube. The desired size of the feeding tube should be determined clinically, and the Gravitas 5Fr Feeding Tube should only be placed if that size is appropriate.

Inclusion Criteria:

* Age at enrollment: 0 to 18 weeks post-partum. Can be up to 12 weeks preterm (gestational age ≥ 28 weeks).
* Suitable to start enteral feeding
* Anticipated to receive enteral feeding (either bolus or continuous feeds) for more than 6 hours and conclude the enteral nutrition while in the care of the NICU. If enteral nutrition has already been initiated, indicated for replacement of an orogastric/nasogastric feeding tube.

Exclusion Criteria:

* Known major upper airway malformation (e.g. tracheoesophageal fistula)
* Known major GI malformation (e.g. malrotation)
* NPO status -neonate expected to remain NPO for the following 72 hours
* Has a medical condition that drastically affects gastric acid-secretion (e.g. Zollinger-Ellison Syndrome, congenital achlorhydria, gastrointestinal perforation/leak/obstruction)
* Has had removal of part of the stomach
* Critically ill, facing imminent death
* Neonate on ECMO
* Deemed unsuitable for enrollment in study by the site principal investigator based on the patients' medical history
* Ability to have a legally authorized representative provide informed consent

Both neonates on a ventilator (non-invasive or invasive ventilation) or not requiring a ventilator are eligible for this study.

Ages: 0 Weeks to 18 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates in NICU
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Percentage of accurate verifications of anatomical locations of the tip of the Gravitas feeding tube. | 5 months
  Data collected during the study will be post processed to refine the Gravitas placement algorithm. The position of the feeding tube tip as processed by the Gravitas placement algorithm will be compared to institutional standard of care.
Percentage of accurate removals/dislodgements identified by the Gravitas dislodgement algorithm. | 5 months
  Data collected during the study will be post processed to refine the Gravitas placement algorithm. The removal/dislodgement of the feeding tube tip as processed by the Gravitas placement algorithm will be compared to actual removal/verification of dislodgement by institutional standard of care.
Adverse events (a) related to placement and (b) throughout the duration of the presence of the feeding tube within the patient. | 5 months
  The number and type of adverse events will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No